CLINICAL TRIAL: NCT03225560
Title: A Novel Smart Phone Application for Patients Undergoing COLOnoscopic Bowel PREParation: A Randomized Controlled Trial
Brief Title: Smart Phone App for COLOnoscopic PREParation
Acronym: COLOPREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunil Patel (Other)
Responsible Party: Sponsor-Investigator, Sunil Patel, Assistant Professor and Attending Surgeon, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6020364
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer Screening; Colonoscopy; Mass Screening
Keywords: Smart Phone Application; Bowel Preparation; Colorectal Cancer Screening
MeSH Terms: interventions — Cathartics

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be aware of the arm they were assigned to. Colonoscopist performing the colonoscopy will be masked to the intervention and will be providing the assessment of the quality of bowel preparation.
  The investigators will be masked to the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Phone Application (Experimental): A novel smart phone application available for both Apple iOS and Google Android platforms with capabilities to populate the phone calendar with automated reminders/notifications at the appropriate times prior to the colonoscopy.
  Interventions: Other: Bowel Preparation
- Traditional Paper Instructions (Active Comparator): Traditional paper instructions for bowel preparation
  Interventions: Other: Bowel Preparation

INTERVENTIONS:
Other: Bowel Preparation — Bowel Preparation is completed prior to colonoscopy to ensure adequate visualization of the bowel lumen. This requires diet modifications and taking of medications at specified time intervals.

SUMMARY:
This is a randomized controlled trial designed to assess the efficacy of a novel smartphone application as an automated reminder tool in improving the quality of bowel preparation for patients undergoing outpatient colonoscopies. The investigators will be comparing the smartphone application to traditional instructions for bowel preparation. The quality of bowel preparation will be assessed using the Ottawa and Aronchick bowel preparation scales.

DETAILED DESCRIPTION:
This is a randomized controlled trial designed to assess the efficacy of a novel smartphone application as an automated reminder tool in improving the quality of bowel preparation for patients undergoing outpatient colonoscopies at an academic teaching hospital in Kingston, Ontario.

The intervention under investigation is the use of a novel smart phone application which serves as an automated reminder system for patients undergoing outpatient colonoscopies. The application requires the patients to enter the date and time of the colonoscopy appointment and automatically populates the patients' phones with calendar reminders as well as pre-recorded messages regarding cessation of solid food intake, the need for clear fluid intake, as well as timing of their bowel regimens starting 7 days prior.

The design of this study is a prospective, randomized controlled trial with single blinding (endoscopist). Eligible participants will be randomized into either the control (routine paper instructions) or the intervention group (smart phone application). Those who are randomized into the intervention group will be provided with specific instructions to download and setup the smart phone application at least 7 days prior to their scheduled appointment. Upon arrival to their appointment, participants in both groups will be asked to complete a survey confirming the adherence to either paper instructions or instructions provided by the smart phone application.

The primary outcome of this study is the adequacy of the bowel preparation, as assessed by using the Ottawa and Aronchick bowel preparation scales, which have been previously validated and are in common usage for colonoscopy procedures. Secondary outcomes include rate of polyp detection, rate of cecal intubation, and patient reported ease of use and adherence to the bowel regimen instructions.

ELIGIBILITY:
Inclusion Criteria:

* Access to smart phone with the ability to download smart phone application
* Outpatient screening colonoscopy

Exclusion Criteria:

* Patient refusal
* Bowel preparation other than pico-salax or GoLytely
* Urgent/Emergent Colonoscopy
* Patient requiring combined upper and lower endoscopic evaluation
* No access to smart phone or inability to download smart phone application
* Surveillance colonoscopy for previously resected cancer
* Inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Quality of Bowel Preparation | At time of colonoscopy
  The quality of bowel preparation as assessed by the validated Boston and Aronchick bowel preparation scales

SECONDARY OUTCOMES:
Cecal Intubation | At time of colonoscopy
  The ability for the colonoscopist to intubate the cecum
Adenomatous polyp detection | At time of colonoscopy
  The number of adenomatous polyps detected
Patient reported adherence to bowel preparation instructions | At time of colonoscopy
  Patient questionnaire used to determine the adherence to the pre-specified bowel preparation instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil V Patel, MD MSc, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided